CLINICAL TRIAL: NCT06827431
Title: Efficacy and Safety of Ammoxetine Hydrochloride Enteric-coated Tablets in Subjects With Depression: A Multicenter, Randomized, Double-blind, Double-Dummy, Placebo-controlled and Sertraline Active-controlled, Parallel-group, Phase III Study
Brief Title: The Research of Ammoxetine Hydrochloride Enteric-coated Tablets in Subjects With Depression
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: CSPC ZhongQi Pharmaceutical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HA1406-007
Record Dates: First submitted 2024-12-30; First posted 2025-02-14 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2024-12

CONDITIONS: Major Depressive Disorder (MDD)
MeSH Terms: conditions — Depressive Disorder, Major | interventions — ammoxetine; Sertraline

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Ammoxetine group-cohort 1 (Experimental): The eligible subjects will receive Ammoxetine plus placebo.
  Interventions: Drug: Ammoxetine
- Ammoxetine group-cohort 2 (Experimental): The eligible subjects will receive Ammoxetine plus placebo.
  Interventions: Drug: Ammoxetine
- Placebo group (Placebo Comparator): The eligible subjects will receive placebo.
  Interventions: Drug: Placebo
- Sertraline group (Active Comparator): The eligible subjects will receive Sertraline plus placebo.
  Interventions: Drug: Sertraline

INTERVENTIONS:
Drug: Ammoxetine — Drug: Ammoxetine Ammoxetine hydrochloride enteric-coated tablets Drug: Placebo placebo to Ammoxetine and Sertraline.
  Arms: Ammoxetine group-cohort 1
Drug: Ammoxetine — Drug: Ammoxetine Ammoxetine hydrochloride enteric-coated tablets Drug: Placebo placebo to Sertraline.
  Arms: Ammoxetine group-cohort 2
Drug: Placebo — Drug: Placebo placebo to Ammoxetine hydrochlorid and Sertraline.
  Arms: Placebo group
Drug: Sertraline — Drug: Sertraline positive control Drug: Placebo placebo to Ammoxetine hydrochlorid.
  Arms: Sertraline group

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of Ammoxetine hydrochloride enteric-coated tablets in subjects with depression.

DETAILED DESCRIPTION:
In this study, a randomized, double-blind, double-dummy, placebo-controlled and Sertraline active-controlled multicenter study will be conducted to evaluate the efficacy and safety of different doses of Ammoxetine hydrochloride enteric coated tablets in the treatment of depression.

ELIGIBILITY:
Inclusion Criteria:

* 1. Subjects aged 18 and 65 years (inclusive), no gender limitation;
* 2. Subject has recurrent Major Depressive Disorder (MDD) as the primary diagnosis according to Diagnostic and Statistical Manual of Mental Disorders (DSM-5, 5th Edition), single episode or recurrent episodes (classification code 296.2/296.3).The duration of the current depressive episode should be ≥3 months for first-episode patients and ≥1 month for relapsing patients;
* 3. Subjects with a Montgomery-Asberg Depression Rating Scale (MADRS) score ≥ 26 at screening and baseline. Subjects with Clinical Global Impression Scale Disease Severity CGI-S severity score ≥ 4 at screening and baseline. Score of first item (depressed mood) of the HAMD-17 scale ≥2 at the screening and baseline.
* Be able to read and understand the study procedures and trial requirements, agree to abide by the restrictions of the trial and return to the site on time for evaluation, and sign the informed consent form prior to the trial.

Exclusion Criteria:

* 1. Subjects with ≥ 25% reduction in MADRS score in the baseline period compared to the screening period;
* 2. There is a clinically significant risk of suicide or risk of self-injury and harm to others. Those who meet any of the following:

  1. A score of ≥4 on item 10 (Suicidal Ideation) of the MADRS scale;
  2. Subjects who in the judgment of the investigator, are at significant risk for suicide (e.g., participant answered "yes" to question 4 (active suicidal ideation with intent to act but no specific plan) or question 5 (active suicidal ideation with a specific plan and intent) on the Screening C-SSRS and the most recent suicidal intent or suicidal plan occurred within the last six months);
  3. Attempted suicide during the current depressive episode;
* 3. Subjects meet DSM-5 diagnostic criteria for other mental disorders (Schizophrenia spectrum and other psychotic disorders, bipolar and related disorders, anxiety disorders, obsessive-compulsive and related disorders, somatic symptoms and related disorders, substance-related and addiction disorders, etc.)
* 4. Subjects who meet any of the following diagnoses of depressive disorders:

  1. Those who have been determined by the investigator to have TRD (current or prior use of 2 or more antidepressants with different mechanisms that have not been effective with a full course (at least 8 weeks) of treatment at the full dosage (the maximum recommended amount of the instructions);
  2. Subjects with depressive disorders due to other types of mental disorders or somatic diseases (e.g., depressive disorders due to hypothyroidism);
  3. Subjects with depressive disorders due to substances/drugs;
* 5. Subjects who stopped using the following drugs for less than 5 half-lives prior to randomization:

  1. CYP2C19 and CYP3A4 strong inducers and strong inhibitors (e.g., fluoxetine, rifampicin, carbamazepine, etc.);
  2. Combined use of drugs that cause QTc interval prolongation (e.g., levofloxacin, fluconazole, ondansetron, amiodarone, metronidazole, erythromycin, and haloperidol, etc.) or drugs that can cause QTc interval prolongation and may induce torsade de pointes ventricular tachycardia;
  3. Antipsychotics, antidepressants, or mood stabilizers;
* 6. Subjects who have failed previous treatment with a full course (at least 8 weeks) of sertraline at the maximum recommended dose or who have a known allergy to sertraline;
* 7. Subjects who stopped using MAOI (e.g., phenelzine, isocarbazide, antiphencyclidine, linezolid, methylene blue, etc.) for less than 2 weeks before randomization;
* 8. Subjects on long half-life antipsychotics;
* 9. Subjects who have received any of the following non-pharmacologic treatments within 3 months prior to screening:

  1. Electroconvulsive therapy (ECT)
  2. Systemic psychotherapy (e.g., interpersonal therapy, motivational therapy, cognitive behavioral therapy, etc.)
  3. Transcranial magnetic stimulation therapy (TMS)
  4. Vagus Nerve Stimulation (VNS)
  5. Light therapy, etc.
  6. Or those who, in the judgment of the investigator, currently require the above treatments
* 10. Participation in any clinical trial within 3 months prior to screening;
* 11. Those with degree II or III AV block, long QT syndrome, or QTcF >450 ms (males)/460 ms (females) on 12-lead ECG at the time of screening, or those deemed unsuitable for enrollment by the investigator (e.g., tachyarrhythmias requiring clinical management, etc.)
* 12. Screening subjects with ALT or AST greater than 2 times the upper limit of laboratory normal; Severe subclinical hypothyroidism (thyroid function indices only with abnormally elevated TSH and TSH ≥ 10.0 mIU/L); Abnormalities in 2 or more of the 5 thyroid function parameters (TSH, FT3, FT4, TT3, or TT4 values less than 0.9 times the lower limit of normal or more than 1.1 times the upper limit of normal);
* 13. Allergic constitution (e.g. allergic to two or more drugs or to SNRIs);
* 14. Prior history of seizures; or any other condition that increases the risk of seizures (e.g., stroke, severe head trauma, significant metabolic disorders, etc.);
* 15. By the judgment of the investigator, presence of any clinically significant hematologic, endocrine/metabolic, cardiovascular, respiratory, renal, hepatic, gastrointestinal, infectious, or neurological disease or the presence of an unstable or progressive chronic disease that unsuitable for entry into the study;
* 16. History of malignancy, including solid tumors, hematologic malignancies, and carcinoma in situ (except completely resected and cured basal cell carcinoma of the skin, squamous cell carcinoma, and carcinoma in situ of the cervix), within 5 years prior to screening;
* 17. Previous history of increased intraocular pressure or narrow-angle glaucoma;
* 18. Subjects with conditions that interfere with the absorption of oral medications, such as active enteropathy, partial or complete intestinal obstruction, and chronic diarrhea, etc;
* 19. Female subjects who are breastfeeding or have a positive pregnancy test during the screening period or during the study;
* 20. Alcohol or drug dependence within 3 months before screening;
* 21. Male or female with fertility do not agree to use an effective method of contraception during the study and for 1 month after the end of the trial to ensure that contraception is effective for the sexual partner or for themselves;
* 22. Subjects who in the opinion of the investigator, have any other condition that makes them unsuitable for participation in this trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 770 (Estimated)
Dates: Start 2025-02-14 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in Montgomery Asperger Depression Scale (MADRS) score at the end of treatment (week 8) | From baseline to Week 8
  The MADRS is a clinician-rated scale to assess depressive symptomatology during the preceding week. Participants are rated on 10 items (feelings of sadness, lassitude, pessimism, inner tension, suicidality, reduced sleep or appetite, difficulty concentrating, and lack of interest) each on a 7-point scale from 0 (no symptoms) to 6 (symptoms of maximum severity). The total score ranges from 0 to 60 with a higher score indicating more depression. A negative change score indicates improvement

SECONDARY OUTCOMES:
Change from baseline in Hamilton Depression Scale (HAMD-17) at the end of treatment (week 8) | From baseline to Week 8
  The HAMD-17 is a clinician-based assessment of depressive symptoms. The total score ranges from 0 to 53 with a higher score indicating more depression. A score of 0-9 is generally accepted to be within the normal range (or in clinical remission), while a score of greater than 17 indicates moderate to severe depression symptoms.
Change from baseline in The Clinical Global Impression Scale (CGI-S) scores at the end of treatment (week 8) at the end of treatment (week 8) | From baseline to Week 8
  The CGI-S evaluates the severity of psychopathology on a scale of 0 to 7. Considering total clinical experience, a participant is assessed on severity of mental illness at the time of rating according to: 0=not assessed; 1=normal (not at all ill); 2=borderline mentally ill; 3=mildly ill; 4=moderately ill; 5=markedly ill; 6=severely ill; 7=among the most extremely ill participants. The CGI-S permits a global evaluation of the participant's condition at a given time.
Clinical Global Impression Scale of Improvement (CGI-I) score at the end of treatment (week 8) | Week 8
  The CGI-I scale is a clinician-rated instrument that measures the improvement of the participant's symptoms of depression. It is a 7-point scale where a score of 1 indicates that the participant is "very much improved," a score of 4 indicates that the participant has experienced "no change," and a score of 7 indicates that the participant is "very much worse."
The efficiency and remission of the MADRS score | Baseline and week 8
  Effectiveness is defined as ≥ 50% reduction in MADRS score relative to baseline after treatment. Remission is defined as MADRS score ≤ 10 after treatment.
The efficiency and remission of the HAMD-17 score | Baseline and week 8
  Effectiveness is defined as ≥50% reduction in HAMD-17 score relative to baseline after treatment. Remission is defined as HAMD-17 score ≤7 after treatment.
CGI-I score | Week 1, week 2, week 4 and week 6
  The CGI-I scale is a clinician-rated instrument that measures the improvement of the participant's symptoms of depression. It is a 7-point scale where a score of 1 indicates that the participant is "very much improved," a score of 4 indicates that the participant has experienced "no change," and a score of 7 indicates that the participant is "very much worse."
Change from baseline in HAMD-17 score | Week 1, week 2, week 4 and week 6
  The HAMD-17 is a clinician-based assessment of depressive symptoms. The total score ranges from 0 to 53 with a higher score indicating more depression. A score of 0-9 is generally accepted to be within the normal range (or in clinical remission), while a score of greater than 17 indicates moderate to severe depression symptoms.
Change from baseline in MADRS score | Week 1, week 2, week 4 and week 6
  The MADRS is a clinician-rated scale to assess depressive symptomatology during the preceding week. Participants are rated on 10 items (feelings of sadness, lassitude, pessimism, inner tension, suicidality, reduced sleep or appetite, difficulty concentrating, and lack of interest) each on a 7-point scale from 0 (no symptoms) to 6 (symptoms of maximum severity). The total score ranges from 0 to 60 with a higher score indicating more depression. A negative change score indicates improvement.
Change from baseline in HAMA score | Week 1, week 2, week 4 and week 6
  The HAMA is a clinician-rated instrument administered to assess severity of anxiety, its improvement during the course of treatment, and the timing of such improvement. This instrument will be completed by qualified and trained Investigator site raters based on a semi-structured interview for his/her assessment of the participant. The scale consists of 14 items. Each item is rated on a scale of 0 (feeling not present) to 4 (very severe prevalence of the feeling). The HAMA total score is the sum of the 14 items and the score ranges from 0 to 56.
Change from baseline in CGI-S score | Week 1, week 2, week 4 and week 6
  The CGI-S evaluates the severity of psychopathology on a scale of 0 to 7. Considering total clinical experience, a participant is assessed on severity of mental illness at the time of rating according to: 0=not assessed; 1=normal (not at all ill); 2=borderline mentally ill; 3=mildly ill; 4=moderately ill; 5=markedly ill; 6=severely ill; 7=among the most extremely ill participants. The CGI-S permits a global evaluation of the participant's condition at a given time.
The efficiency and remission of the HAMD-17 score | Week 1, week 2, week 4 and week 6
  Effectiveness is defined as ≥50% reduction in HAMD-17 score relative to baseline after treatment. Remission is defined as HAMD-17 score ≤7 after treatment.
The efficiency and remission of the MADRS score | Week 1, week 2, week 4 and week 6
  Effectiveness is defined as ≥ 50% reduction in MADRS score relative to baseline after treatment. Remission is defined as MADRS score ≤ 10 after treatment.
The percentage of subjects with a MARDS score reduction ≥ 25% | Week 1and week 2

IPD SHARING:
Plan to Share IPD: No